CLINICAL TRIAL: NCT02753335
Title: A Randomized Trial of Patients With Complex Regional Pain Syndrome Comparing Graded Motor Imagery and Desensitization Versus Simple Desensitization and Changes in Resting-State Connectivity of Cerebral Networks Before and After Treatment.
Brief Title: A Comparison of Two Treatments for CRPS and Changes in Resting-State Connectivity of Cerebral Networks.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Tromso (Other)
Collaborators: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2014/1671(REK)
Record Dates: First submitted 2016-03-03; First posted 2016-04-27 (Estimated); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Complex Regional Pain Syndrome
Keywords: CRPS, graded motor imagery, desensitization, fMRI, DMN
MeSH Terms: conditions — Complex Regional Pain Syndromes | interventions — Desensitization, Psychologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GMI and Desensitization (Experimental): Left/right judgement, imagine movements of the affected area, mirror treatment and tactile stimulation of the affected limb with different materials.
  Interventions: Behavioral: GMI and Desensitization
- Desensitization (Experimental): Tactile stimulation of the affected limb with different materials.
  Interventions: Behavioral: Desensitization

INTERVENTIONS:
Behavioral: GMI and Desensitization — Graded Motor Imagery (GMI) is used to treat chronic pain conditions and movement problems related to alterations in the nervous system such as CRPS, postamputation limb pain and back pain. The patient is trained in monitored steps. The three treatment components include left/right discrimination training, motor imagery exercises and mirror observations of the unaffected limb, appearing as the affected limb. They are performed sequentially, but require a flexible approach to suit the individual patient. The imagined movements have been demonstrated to activate motor cortical areas similar to those activated in the actual execution of that movement.
  Desensitization (D) is used to decrease hyperalgesia by repeated tactile stimulation of the affected area with various materials.
  Arms: GMI and Desensitization
Behavioral: Desensitization — Desensitization (D) is used to decrease hyperalgesia and allodynia by repeated tactile stimulation of the affected area with various materials.
  Arms: Desensitization

SUMMARY:
The intention of this trial is to investigate whether combined Graded Motor Imagery (GMI) and Desensitization (D) among patients with CRPS is clinically more effective than only D and to study changes in connectivity in the Default Mode Network before and after treatment.

DETAILED DESCRIPTION:
CRPS: Complex regional pain syndrome (CRPS) is characterized by severe and disabling pain typically in a limb in combination with sensory, autonomic, trophic, and motor abnormalities like tremor and dystonia. A distinction is made between CRPS-1, usually following an injury (fracture, surgery) without a nerve lesion, and CRPS-2, in which a distinct nerve lesion can be identified.

Brain mapping studies have provided increasing evidence that the central nervous system is playing an important role in the pathogenesis of CRPS. Reorganization of the somatosensory cortex and motor networks, with altered central processing of tactile and nociceptive stimuli as well as movement control has been demonstrated.

Functional brain imaging studies suggest that the volume of brain activation differs between motor execution and motor imagery, but the distribution of cerebral activity tends to be similar. Under imaginary movement of affected hands Gieteling et al. (2008) observed that there was reduced activation ipsilaterally in the premotor and adjacent prefrontal cortex, frontal operculum, anterior part of the insula cortex, and the superior temporal gyrus.

Stimulus-driven, functional magnetic resonance imaging, however, are time-consuming and prone to possible confounds, especially in clinical populations. In that perspective resting-state functional magnetic resonance imaging (RS-fMRI), measuring the cerebral networks at rest (in absence of any task), is probably better suited to clinical examinations and is widely used to investigate brain networks that exhibit correlated fluctuations. During recent years, a large number of studies have indicated that RS-fMRI is sufficiently constrained by anatomy to allow the architecture of distinct brain systems to be characterized.

The default mode network (DMN) is probably the most studied resting state network. It seems to be involved in several processes and is found negatively modulated by chronic pain. Only one published study has investigated cerebral networks and cerebral connectivity in CRPS. Here the default mode network displayed reduced connectivity with the S1 compared to healthy controls. This indicates that decreased connectivity may be a key feature in cerebral functioning of CRPS patients. No study, however, has so far investigated if the reduced connectivity in the DMN is reversed in CRPS patients who experience pain reduction after GMI or desensitization treatment.

Diffusion tensor imaging (DTI) is another magnetic resonance technique useful for revealing microstructural properties of tissue, particularly in cerebral white matter.

Chronic pain has also been associated with reduced cognitive functioning. If this is caused by pain processing demands, competing with working memory and executive functions, the investigators would expect the cognitive capacity to be improved or restored if the pain is successfully treated.

Graded Motor Imagery: Graded Motor Imagery (GMI) is a rehabilitation process and has been used to treat chronic pain conditions and movement problems related to alterations in the nervous system such as CRPS, postamputation limb pain, and back pain. The patients are trained in monitored steps which increase in difficulty as progress is made. The three treatment components include left/right discrimination training, motor imagery exercises and mirror observations of the unaffected limb, appearing as the affected limb. The components are performed sequentially, but require a flexible approach to suit the individual patient. The imagined movements have been demonstrated to activate motor cortical areas similar to those activated in the actual execution of that movement.

Desensitization: Tactile desensitization (D) is used to decrease hyperalgesia and allodynia by repeatedly touching the affected area with various materials. This has successfully been used clinically in the treatment of CRPS.

Hypotheses: The following hypotheses will be investigated:

1. Patients, treated with GMI + D, experience a larger pain reduction compared with those subjected to D only.
2. Non-responders to D alone experience pain reduction when D is combined with GMI.
3. Patients with CRPS display reduced intra-network connectivity in the DMN compared to healthy controls.
4. Reduced intra-network connectivity in CRPS is associated with pain intensity.
5. Reduced connectivity in the DMN is reversed in patients who experience pain reduction after GMI and D treatment. This will be evident in the comparison of fMRI data obtained before and after treatment.
6. Microstructure of the cerebral white matter is changed during the intervention.

Design:The effects of treatment with Graded Motor Imagery (GMI ) and D versus D alone will be compared with an open, randomized, semi-cross-over case-control design.

The study patients will be allocated to either GMI+D or D alone. After an initial treatment period of six weeks responders (R) stay in the same treatment group and continue this treatment. Non-responders (NR) in the D treatment group will be offered an immediate combined treatment (GMI+D).

Randomization: The recruited patients will be allocated in a ratio 1:1 by randomization with a fixed block size of 6.

Analytical models: Self reported symptom burden and functional capacity will be compared between the two treatment groups and within each treatment group (i.e. comparisons before and after treatment and with each patient as his/her own control).

The investigators will also compare the two intervention groups (CRPS patients receiving a GMI+D and D alone) with a non-randomized comparison group of sex- and age-matched healthy persons.

Continuous, symmetrically distributed variables will be expressed by mean values with 95% confidence intervals (95% CI) constructed by the Student procedure. Proportions will be presented using the Binomial model with the exact 95% calculated confidence interval.

Assumed continuously distributed variables will be analyzed by Analysis of Variance (ANOVA) model with the initial value as covariate while contingency table analysis is used for group comparisons of categorical and ranked variables.

The sample size calculation is based on distribution of the main variable, self-rated limb pain measured by Visual Analogue scaling (VAS). Based on the assumption of normality, a significance level of 5 % (α = 0.05), a power of (β = 0.80) and a clinical relevant difference of one time Standard Deviation (SD), 21 patients should be included in each of the two treatment groups. There will also be a sex- and age-matched comparison group of healthy persons (n:21).

Interventions:

Individually adjusted Graded motor imagery (GMI) and tactile desensitization (D).

Measurements:

MRI-scanning (for analyses of Intra-network connectivity in the DMN and DTI for microstructural changes in the white matter), Quantitative Sensory Testing (QST) and Neuropsychological tests are performed before the randomization and 12 months later.

Self reporting questionnaires will be performed at baseline, after the treatment period of six weeks, and at the 6 and 12 month follow up.

This includes demographic variables, and a comorbidity check list of diseases related to the major organ systems, pain intensity measured by numerical scales for pain intensity and by Visual Analogue Scale (VAS), consumption of analgesics and the questionnaires: CRPS Severity Score, if upper limb affected; Quick DASH (a short form of Disabilities of the Arm, Shoulder and Hand Outcome Measure), if lower limb affected; Lower extremity functional scale, Impact of Event Scale-6 if subjected to adverse life events, Insomnia Severity Index, The Hopkins Symptoms Checklist (HSCL- 25), Pain Catastrophizing Scale, Perceived self efficacy and the Bath CRPS Body Perception Disturbance Scale

ELIGIBILITY:
Inclusion criteria:

* Patients 18 - 70 years old. For patients who only participate in the clinical RCT (without fMRI) no upper age limit.
* CRPS affecting one single upper or lower limb diagnosed by the IASP (2012) Budapest research criteria (Harden et al., 2010).
* Triggering trauma or the onset of pain >3 months ago.
* If possible drugs that can influence the fMRI scans should be avoided. Documentation if used.

Exclusion criteria

* Drug abuse.
* Malignant/progressive, systemic or neurodegenerative disease.
* Other severe pain conditions.
* Severe clinical anxiety or depression, symptoms of fatigue or ME of a disabling level.

For patients who participate in the MRI related analyses:

* Metallic implants incompatible with the MR technology or medical condition not recommended for fMRI.
* Pregnancy.
* Phobia for MRI examination.
* Diseases that can cause structural changes and interfere with the interpretation of the MRI-scans (like severe diabetes mellitus, heart disease, ischemic stroke and vascular conditions).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2016-09; Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Group difference in pain intensity | 6 weeks after baseline
  Continuous numeric variable using a visual analog scale from minimum 0 to maximum 100
Change from baseline in intra-network connectivity in the Default Mode Network | 6 months after baseline
  Continuous variable

SECONDARY OUTCOMES:
Change from baseline in pain intensity | 6 weeks after baseline
  Continuous numeric variable using a visual analog scale from minimum 0 to maximum 100
Change from baseline in pain intensity | 6 months after baseline
  Continuous numeric variable using a visual analog scale from minimum 0 to maximum 100
Change from baseline in pain intensity | 12 months after baseline
  Continuous numeric variable using a visual analog scale from minimum 0 to maximum 100
Group difference in CRPS Severity Score | 6 weeks after baseline
  Continuous variable using a numeric scale from minimum 0 to maximum 17
Change from baseline in CRPS Severity Score | 6 weeks after baseline
  Continuous variable using a numeric scale from minimum 0 to maximum 17
Change from baseline in CRPS Severity Score | 6 months after baseline
  Continuous variable using a numeric scale from minimum 0 to maximum 17
Change from baseline in CRPS Severity Score | 12 months after baseline
  Continuous variable using a numeric scale from minimum 0 to maximum 17
Group difference in Quick DASH score/percent lower extremity functional scale score | 6 weeks after baseline
  Continous variable using a numeric scale from minimum 0 to maximum 100
Relative change from baseline in Quick DASH/Lower extremity functional scale score | 6 weeks after baseline
  Continous variable using scales from minimum 0 to maximum 100
Relative change from baseline in Quick DASH/Lower extremity functional scale score | 6 months after baseline
  Continous variable using scales from minimum 0 to maximum 100
Relative change from baseline in Quick DASH/Lower extremity functional scale score | 12 months after baseline
  Continous variable using scales from minimum 0 to maximum 100
Group difference in responder rate | 6 weeks after baseline
  Categorical variable indicating the proportion of patients who reaches a clinically meaningful change (33 % pain reduction) on a numeric rating scale (0-10).
Change from baseline in responder rate | 6 weeks after baseline
  Categorical variable indicating the proportion of patients who reaches a clinically meaningful change (33 % pain reduction) on a numeric rating scale (0-10).
Change from baseline in responder rate | 6 months after baseline
  Categorical variable indicating the proportion of patients who reaches a clinically meaningful change (33 % pain reduction) on a numeric rating scale (0-10).
Change from baseline in responder rate | 12 months after baseline
  Categorical variable indicating the proportion of patients who reaches a clinically meaningful change (33 % pain reduction) on a numeric rating scale (0-10).

CONTACTS AND LOCATIONS:
Overall Officials: Gunnvald Kvarstein, PhD, Study Chair — University of Tromso
Locations (1):
- University Hospital of North Norway, Tromsø, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smart KM, Ferraro MC, Wand BM, O'Connell NE. Physiotherapy for pain and disability in adults with complex regional pain syndrome (CRPS) types I and II. Cochrane Database Syst Rev. 2022 May 17;5(5):CD010853. doi: 10.1002/14651858.CD010853.pub3. PMID 35579382